CLINICAL TRIAL: NCT05547958
Title: Parents InformaTion in Child REHABilitation
Acronym: PITChREHAB
Status: Completed | Type: Observational
Sponsor: Fondation Ildys (Other)
Collaborators: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: IS-C4-2022-009
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Children with Chronic Condition
Keywords: m-health; mobile apps; chronic disease; informations; parents; pediatric; rehabilitation; communication
MeSH Terms: conditions — Chronic Disease; Communication | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Focus group and online survey — Focus group with parents of children with disabilities or chronic condition will be organized to identify hypotheses regarding their needs in terms of informations exchange with pediatric rehabilitation professionals about the rehabilitation care of their children.
  Then, an online survey will be proposed to parents of children with disabilities or chronic condition in France to identify their needs regarding the development of apps that offer the feature to share informations with rehabilitation professionals.

SUMMARY:
In France, approximaly 3 million children have a chronic disease and require regular care such as paediatric rehabilitation. These cares are provided over long periods of time, most often throughout childhood and often into adulthood. Paediatric rehabilitation care involves multidisciplinary team working closely with families. During follow-up rehabilitation, communication between the children, families and the professionals is essential. To this end, digital health solutions can be helpful.

Digital health solutions are rapidly emerging in the field of paediatric rehabilitation. In this context of emergence of digital health solutions, it is essential to identify the needs and expectations of families of children with a chronic disease.

This project aims to identify the key points in terms of information exchange on rehabilitation monitoring. To identify these needs, a mixed study will be carried out from June 2022 to June 2023 involving focus groups to gather qualitative informations on parent's needs in terms of information exchange through digital apps and quantitative research with a survey that will allow to prioritise these needs.

DETAILED DESCRIPTION:
For the first part of the study, the researchers will conduct focus groups and interview parents about their experiences and perceptions of information exchange with rehabilitation professionals. All the participants will be parents of a child with a chronic disease, aged between 0 and 18 years and receiving paediatric rehabilitation care. The objective of this first part is to collect qualitative information on the needs of parents in terms of information exchange through digital applications.

With the analysis of the focus group, the researchers will define the hypothesis.

Then, a survey will be built and shared online in France during 3 months (2nd semester 2022).

With this survey, the objective is to identify the key points for the development of paediatric rehabilitation apps in terms of information exchange.

Quantitative data will be described with frequency, mean and standard deviation.

ELIGIBILITY:
Inclusion Criteria:

- parents of a child (0-18 years) with a chronic condition and with a rehabiilitation follow up

Exclusion Criteria:

* parents who do not speak french
* parents with an intellectual disability (for the first part : focus group)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents of a child (0-18 years) with a chronic condition and with a rehabilitation follow up will be invited by physicians in three pediatric rehabilitation centers to participate to the focus groups.
  The survey will be adressed nationally to the parents of children with a chronic condition and with a rehabilitation follow up.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
key elements desired by parents in the apps aiming to share informations with rehabilitation professionals | june 2022 - june 2023
  The aim is to identify the key priority elements for parents in the design of mobile apps for information exchange with rehabilitation professionals.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ildys, Brest, France

REFERENCES:
- [Background] Nussbaum R, Kelly C, Quinby E, Mac A, Parmanto B, Dicianno BE. Systematic Review of Mobile Health Applications in Rehabilitation. Arch Phys Med Rehabil. 2019 Jan;100(1):115-127. doi: 10.1016/j.apmr.2018.07.439. Epub 2018 Aug 29. PMID 30171827
- [Background] Maguire M. Methods to support human-centred design. International Journal of Human-Computer Studies. 1 oct 2001;55(4):587-634.
- [Background] O'Cathain A, Murphy E, Nicholl J. Three techniques for integrating data in mixed methods studies. BMJ. 2010 Sep 17;341:c4587. doi: 10.1136/bmj.c4587. No abstract available. PMID 20851841
- [Background] de Jongh T, Gurol-Urganci I, Vodopivec-Jamsek V, Car J, Atun R. Mobile phone messaging for facilitating self-management of long-term illnesses. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD007459. doi: 10.1002/14651858.CD007459.pub2. PMID 23235644